CLINICAL TRIAL: NCT05672732
Title: In Depth Observational Clinical Trial Assessing Experiences of Alzheimer's Disease Patients To Determine Trial Attributes Affecting Completion Rates For Specific Demographic Groups
Brief Title: Assessment of Clinical Trial Experiences of Alzheimer's Disease Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 81466128
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Alzheimer's
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Taking part in medical trials usually favors a particular demographic group. But there is limited research available to explain what trial attributes affect the completion of these specific demographic groups.

This study will admit a wide range of data on the clinical trial experience of Alzheimer's Disease patients to determine which factors prevail in limiting a patient's ability to join or finish a trial.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future Alzheimer's Disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 50 to 80 years of age
* Participant has a diagnosis of Alzheimer's Disease
* Patient has self-identified as planning to enroll in an interventional clinical trial for Alzheimer's Disease

Exclusion Criteria:

* No diagnosis of Alzheimer's Disease confirmed
* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Alzheimer's Disease patients who are actively considering involvement in an interventional clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a Alzheimer's Disease Clinical Trial | 3 months
Number of patients who remain in Alzheimer's Disease clinical trial until completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eratne D, Loi SM, Farrand S, Kelso W, Velakoulis D, Looi JC. Alzheimer's disease: clinical update on epidemiology, pathophysiology and diagnosis. Australas Psychiatry. 2018 Aug;26(4):347-357. doi: 10.1177/1039856218762308. Epub 2018 Apr 3. PMID 29614878
- [Background] Mangialasche F, Solomon A, Winblad B, Mecocci P, Kivipelto M. Alzheimer's disease: clinical trials and drug development. Lancet Neurol. 2010 Jul;9(7):702-16. doi: 10.1016/S1474-4422(10)70119-8. PMID 20610346
- [Background] Rafii MS, Aisen PS. Alzheimer's Disease Clinical Trials: Moving Toward Successful Prevention. CNS Drugs. 2019 Feb;33(2):99-106. doi: 10.1007/s40263-018-0598-1. PMID 30560544

DOCUMENTS (1):
  • Informed Consent Form (2023-01-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT05672732/ICF_000.pdf